CLINICAL TRIAL: NCT03925194
Title: A Phase IIa, Randomized, Placebo-controlled, Double-blind, Cross-over Study to Evaluate Safety and Efficacy of Subcutaneous Administration of Anakinra in Patients With Cystic Fibrosis
Brief Title: A Study to Evaluate Safety and Efficacy of Subcutaneous Administration of Anakinra in Patients With CF
Acronym: ANAKIN
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Heidelberg University (Other)
Responsible Party: Principal Investigator, Mirjam Stahl, Deputy of Principal Investigator (Olaf Sommerburg), Heidelberg University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EudraCT No.: 2016-004786-80-A
Record Dates: First submitted 2019-04-19; First posted 2019-04-24 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Cystic Fibrosis, 10011762
MeSH Terms: conditions — Cystic Fibrosis | interventions — Interleukin 1 Receptor Antagonist Protein

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Anakinra (Experimental)
  Interventions: Drug: Anakinra
- Placebo (Placebo Comparator)
  Interventions: Drug: Anakinra

INTERVENTIONS:
Drug: Anakinra — Application of Anakinra once daily for 28 days

SUMMARY:
OBJECTIVES

Primary:

To evaluate efficacy of treatment with anakinra in subjects with CF who are ≥ 12 years of age by means of lung clearance index (LCI).

Secondary To evaluate safety and tolerability of treatment with anakinra as well as to investigate further effects of anakinra on lung function and quality of life (QOL) in subjects with CF.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years (1st cohort). If justified by interim analysis, 18 > age ≥ 12 years (2nd cohort),
2. Informed consent of the patient (if applicable) and/or all legal guardians,
3. Sufficient fluency of patient and/or his/her representative in German language to comply with study-specific procedures (e.g. to complete required quality of life questionnaires),
4. Confirmed diagnosis of cystic fibrosis, fulfilling at least one of the following three criteria:

   1. sweat chloride ≥ 60mEq/L,
   2. two CF causing mutations in the CFTR gene,
   3. alterations of transepithelial potential difference of nasal or rectal epithelia typical for CF,
5. FEV1 ≥ 50 % pred. at screening,
6. LCI2.5 ≥ 7.05 at screening,
7. Ability to perform reproducible multiple breath washout and spirometry,
8. Oxyhaemoglobin saturation of ≥ 90% on room air at screening,
9. No changes in the medication for cystic fibrosis lung disease for at least 4 weeks prior to the first administration of the IMP of each treatment period (in case of medication changes in Period 1 and/or the washout phase the wash-out may be extended for up to 12 weeks in order to fulfill this criterion),
10. Adequate bone marrow function assessed on the basis of: neutrophils >1.5 x 109/L, platelets >100 x 109/L, hemoglobin >9.0 g/dL,
11. Adequate liver function assessed on the basis of: GGT, ASAT, and ALAT <3 x upper limit of normal (ULN),
12. Adequate blood clotting assessed on the basis of: aPTT <39 sec., INR <1.2,
13. Negative serology for HIV (anti-HIV 1/2 IgG/IgM and p24-Ag), HBV (anti-HBs quantitative and anti-HBc IgG/IgM) and HCV (anti-HCV IgG), negative Interferon-gamma release assay,
14. Negative Beta-HCG blood/urine test in women of childbearing potential (of childbearing potential are females who have experienced menarche and are not permanently sterile or postmenopausal (postmenopausal: 12 consecutive months with no menses without an alternative medical cause)),
15. Use of adequate contraception in sexually active female subjects (sexual abstinence, hormonal contraceptives or intrauterine device).

Exclusion Criteria:

1. Expected non-compliance, i.e. inability or unwillingness to comply with study-specific procedures,
2. Known allergy to anakinra or any ingredient of the pharmaceutical formulation of Kineret®,
3. Planned immunization with attenuated (live) vaccine(s) during the treatment with the IMP or completed immunization with attenuated (live) vaccine(s) within 4 weeks prior to the first administration of the IMP,
4. Renal failure (creatinine in serum above ULN),
5. History of tuberculosis or repeated detection of non-tuberculous mycobacteria from airway samples in the last 12 months before start of each treatment period,
6. History of detection of Burkholderia cenocepacia species in the last 12 months before start of each treatment period,
7. Colonization with multi-resistant Staphylococcus aureus (MRSA) and/or 4-multi-resistant gram negative (MRGN) Pseudomonas aeruginosa is only an exclusion criterion if the treating physician judges that this is an increased risk for the patient,
8. Acute bronchopulmonary exacerbation (defined by modified Fuchs criteria (1) (see Appendix 1), modification includes all ways of application of an antibiotic (e.g., oral, i.v., inhaled)) within 14 days prior to the screening and before start of each treatment period,
9. Signs of other active infection within 14 days prior to the screening and before start of each treatment period (clinical symptoms (e.g. burning sensation while urinating, skin, wound or dental infection) and/or fever and/or deterioration of infection-specific laboratory parameters beyond changes driven by the underlying disease),
10. Immunosuppressive treatment due to organ transplantation, rheumatic or autoimmune diseases as well as treatment with Anakinra in the last 3 months before Day 1 of Period 1,
11. Participation in another interventional trial within the last 30 days prior to screening,
12. Current oral corticosteroid use,
13. Current oxygen supplementation,
14. Current treatment with etanercept,
15. Medical history of lung transplantation,
16. Pregnant or nursing females (females of childbearing potential must have a negative pregnancy test at Screening),
17. Known hypersensitivity to hypertonic saline (used for induction of sputum).

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Absolute pre-post change of the lung clearance index (LCI) | 28 days

CONTACTS AND LOCATIONS:
Locations (3):
- Germany (3):
  - University Children's Hospital Heidelberg, Cystic Fibrosis Centre, Heidelberg, Baden-Wurttemberg
  - Universitätsmedizin Essen, Ruhrlandklinik, Essen, North Rhine-Westphalia
  - Charité - Universitätsmedizin Berlin, Berlin, State of Berlin

IPD SHARING:
Plan to Share IPD: No